CLINICAL TRIAL: NCT00091754
Title: Atherosclerosis, Plaque and CVD in Communities
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Eric Boerwinkle, Professor - School of Public Health, The University of Texas Health Science Center, Houston
Other Study IDs: 1269; 5U01HL075572-04 (NIH)
Record Dates: First submitted 2004-09-16; First posted 2004-09-20 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Cerebrovascular Accident; Coronary Arteriosclerosis; Coronary Disease
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Stroke; Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Stored DNA in Atherosclerosis Risk in Communities (ARIC) cohort study to test the ability of the genomic correlates of plaque characteristics to predict incident coronary heart disease and stroke.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify new cellular, metabolic, and genomic correlates of atherosclerotic plaque and early pathologic changes in the vascular wall and determine their consequences for coronary heart disease and stroke.

DETAILED DESCRIPTION:
BACKGROUND:

This study draws upon the existing ARIC cohort of 15,792 members aged 45-64 years at baseline in 1987-1989 who have completed four clinic exams three years apart with the last exam in 1998. The longitudinal ARIC cohort study focused on new cardiovascular disease [CVD] risk factors and subclinical measures of atherosclerosis through B-mode ultrasound of the carotid arteries. The current study collects new and novel risk factors and performs carotid magnetic resonance imaging (MRI) examinations on a stratified random sample of 1,200 ARIC participants with high (>85th percentile) carotid intimal-medial thickness [IMT] by ultrasound and 800 participants with <85th percentile IMT.

DESIGN NARRATIVE:

The study examines an informative subset of the bi-ethnic Atherosclerosis Risk in Communities (ARIC) cohort to identify cellular, metabolic and genomic correlates of atherosclerotic plaque characteristics and of early changes in the vascular wall. The longitudinal follow-up and stored DNA in ARIC will allow testing the ability of the genomic correlates of plaque characteristics to predict incident coronary heart disease and stroke. One thousand two hundred individuals with high (>85th percentile) carotid artery wall thickness documented by B-mode ultrasound and 800 individuals sampled from the remainder of the carotid artery wall thickness distribution (<85th percentile) will receive a contrast-enhanced carotid MRI examination. Standardized MRI measures will include carotid artery wall thickness, T2 signal intensity changes and percent contrast enhancement indicative of endothelial dysfunction, and for those with plaque, fibrous cap thickness, lipid core volume, and calcification. Novel cellular, metabolic and genomic measures will be collected and will be related to MRI-measurable plaque characteristics. In particular, flow cytometry will be used to measure monocyte and platelet presentation of cytokines, growth factors and adhesion molecules, and cell-cell aggregation. High throughput genotyping methods will be used to measure 5 to 7 polymorphic sites in each of 150 positional, expressional and biologic candidate genes, permitting multilocus and haplotype genomic analyses. The depth and breadth of existing risk factor and lifestyle data, extensive follow-up since 1986-89, and accumulation of clinical outcomes, including coronary heart disease, stroke and arteriosclerosis, contribute additional strengths to the laboratory and MRI investigations. Inferences will be made both cross-sectionally and longitudinally, with a special emphasis on genotype plus environment interaction. The ARIC cohort is in an ideal age range for the research because of the frequent and documented occurrence of plaque and the spectrum of clinically relevant stages from plaque initiation to mature fibrosis, calcification and even erosion and near-rupture.

ELIGIBILITY:
No eligibility criteria

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The current study collects new and novel risk factors and performs carotid magnetic resonance imaging (MRI) examinations on a stratified random sample of 1,200 ARIC participants with high (>85th percentile) carotid intimal-medial thickness [IMT] by ultrasound and 800 participants with <85th percentile IMT.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2004-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Boerwinkle, Ph.D, Principal Investigator — University of Texas